CLINICAL TRIAL: NCT04686500
Title: VisionRT-based Deep Inspiration Breath-hold (DIBH) Respiratory Motion Management Strategy, A Pilot Study for Thoracic and Abdominal Tumors Stereotactic Body Radiotherapy
Brief Title: VisionRT-based Deep Inspiration Breath-hold (DIBH) Respiratory Motion Management Strategy, A Pilot Study for Thoracic and Abdominal Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Vision RT Limited (Industry)
Responsible Party: Principal Investigator, David Parsons, PhD, ASSISTANT PROFESSOR, Radiation Oncology - RO-Medical Physics&Engineering, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 022017-075
Record Dates: First submitted 2020-11-30; First posted 2020-12-28 (Actual); Results first posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-10

CONDITIONS: Thoracic Cancer; Abdominal Cancer

STUDY DESIGN:
Intervention Model Description: Prospective study with retrospective data analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Inspiration Breath-hold (DIBH) Respiratory Motion (Other): DIBH qualified patient will experience one high-resolution CT scan as SOC and additional 3 low resolution/lower dose CT scans to further investigate inter-DIBH patient surface and tumor position stability and repeatability
  Interventions: Device: Tidal volume measured by spirometer and DIBH surface from CT image

INTERVENTIONS:
Device: Tidal volume measured by spirometer and DIBH surface from CT image — The SOC DIBH CT scan will be transferred to Eclipse treatment planning system for treatment planning. Tidal volume measured by spirometer and DIBH surface from CT image will be used as a reference surface for patient treatment initial setup. CBCT will be acquired before each fractional treatment for the patient alignment before beam delivery.

SUMMARY:
A more recent competing technology for implementing the DIBH technique is real-time surface photogrammetry using the AlignRT system (Vision RT Ltd., London, UK). AlignRT system use non-ionization near infrared light to track patient surface motion. The system has one projector projecting near infrared optical pattern on patient surface. The optical pattern is imaged by optical cameras (two per pod) at ~25 Hz. The user selects a region-of-interest (ROI) on the surface and the software calculates and displays the real-time position in six degrees (3 translations and 3 rotations) in real-time. Once the patient has matched the pre-determined DIBH position (within threshold accuracy), the radiation beam is enabled to be turned on for treatment.

DETAILED DESCRIPTION:
VRT-DIBH has already applied to left breast radiotherapy to spare lung and heart. Compared to ABC-DIBH, VRT-DIBH has several potential advantages:

1. VRT monitors patient (surface) position in addition to DIBH signal, while ABC only check the tidal volume, which can remain the same even if the patient shifts slightly on the couch;
2. VRT is more cost effective, as patient tubing needs to be replaced daily for ABC;
3. VRT potentially has advantage on patient compliance, as with ABC breath is forced impeded while with VRT breath-hold is voluntary.

In this study, we renovate the established DIBH motion management strategy by adopting AlignRT system. The purpose of this study is to develop, validate, and prove the feasibility of VRT-DIBH technique for lung and liver SBRT.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be willing and capable to provide informed consent to participate in the protocol.
2. Patient with presumed pulmonary function capable of holding breath for at least 30 seconds - later to be confirmed.
3. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, and until study imaging is complete. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

3.1 A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:

* Has not undergone a hysterectomy or bilateral oophorectomy; or
* Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).

3.2 Patients must be compliant to all required pretreatment evaluations

Exclusion Criteria:

1. Pregnant or lactating women, as treatment involves unforeseeable risks to the embryo or fetus
2. Patients are not compliant to all required pretreatment evaluations

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2023-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Parsons, PHD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Deep Inspiration Breath-hold (DIBH) Respiratory Motion
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Deep Inspiration Breath-hold (DIBH) Respiratory Motion
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Correlation Between Kilovoltages X-ray Images of the Diaphragm and the Surface Guided Motion Analyzed With Matlab
Description: VRT-DIBH (VisionRT-based deep inspiration breath-hold) feasibility will be evaluated using descriptive statistics to explore the geometry accuracy and to characterize tumor motion/surface stability and repeatability during treatment. CT images of the treatment site, as well as kV projections and VRT surface images, will be taken and analyzed for this purpose. The trajectory data and kV projection data were analyzed in Matlab. In the kV images, the diaphragm was segmented and used for tracking of the BH position. This was done using several steps including: derivatives, polynomial curve fitting and high pass filtering. The correlation was then measured using a Pearson correlation. Correlation of each breath hold was taken and averaged.
Time Frame: 1 month
Measure: Mean (Full Range); unit: correlation coefficient
Arm/Group | Deep Inspiration Breath-hold (DIBH) Respiratory Motion
Number analyzed (Participants) | 10
correlation coefficient
  Vertical | 0.01 [-0.07 to 0.3]
  Longitudinal | 0.07 [-0.04 to 0.73]

2. Secondary Outcome: Target Margin Contingency Table Based on Surface and Diaphragm Motion
Description: To assess the necessary margin for a target, the amount of surface and diaphragm motion was analyzed. For each x-ray image the diaphragm motion and corresponding surface motion were recorded. These motions were then categorized based on their size and researchers counted how often these movements fell within the specified motion ranges.
Time Frame: 1 month
Population: Outcomes for secondary objectives have been combined in this contingency table between motion range of kV and motion of superior-inferior and anterior-posterior surfaces.
Measure: Number; unit: sample points (number of movements)
Groups:
- Bin [0 1)mm kV; Bin [1 2)mm kV; Bin [2 3)mm kV; Bin [3 4)mm kV; Bin [4 5)mm kV; Bin [5 10)mm kV: Contingency table motion range for kV
- Total kV: Contingency table totals
Arm/Group | Bin [0 1)mm kV | Bin [1 2)mm kV | Bin [2 3)mm kV | Bin [3 4)mm kV | Bin [4 5)mm kV | Bin [5 10)mm kV | Total kV
Number analyzed (Participants) | 10 | 10 | 10 | 10 | 10 | 10 | 10
sample points (number of movements)
  Bin [0 1)mm (Superior-Inferior Motion) | 16172 | 2161 | 428 | 92 | 26 | 14 | 18893
  Bin [1 2)mm (Superior-Inferior Motion) | 3844 | 741 | 248 | 50 | 12 | 7 | 4902
  Bin [2 3)mm (Superior-Inferior Motion) | 1082 | 257 | 102 | 26 | 10 | 9 | 1486
  Bin [3 4)mm (Superior-Inferior Motion) | 506 | 105 | 24 | 9 | 4 | 2 | 650
  Bin [4 5)mm (Superior-Inferior Motion) | 216 | 44 | 11 | 2 | 1 | 2 | 276
  Bin [5 10)mm (Superior-Inferior Motion) | 304 | 52 | 13 | 3 | 0 | 0 | 372
  Bin [10 15)mm (Superior-Inferior Motion) | 19 | 5 | 3 | 0 | 0 | 0 | 27
  Bin [15 20)mm (Superior-Inferior Motion) | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Total (Superior-Inferior Motion) | 22143 | 3365 | 829 | 183 | 53 | 34 | 26607
  Bin [0 1)mm (Anterior-Posterior Motion) | 19344 | 2846 | 711 | 157 | 48 | 28 | 23134
  Bin [1 2)mm (Anterior-Posterior Motion) | 1798 | 288 | 59 | 21 | 4 | 3 | 2173
  Bin [2 3)mm (Anterior-Posterior Motion) | 493 | 106 | 18 | 5 | 1 | 3 | 626
  Bin [3 4)mm (Anterior-Posterior Motion) | 181 | 38 | 7 | 0 | 0 | 0 | 226
  Bin [4 5)mm (Anterior-Posterior Motion) | 97 | 21 | 3 | 0 | 0 | 0 | 121
  Bin [5 10)mm (Anterior-Posterior Motion) | 192 | 54 | 28 | 0 | 0 | 0 | 274
  Bin [10 15)mm (Anterior-Posterior Motion) | 38 | 12 | 3 | 0 | 0 | 0 | 53
  Total (Anterior-Posterior Motion) | 22143 | 3365 | 829 | 183 | 53 | 34 | 26607

ADVERSE EVENTS:
Time Frame: AEs were not collected for this trial
Description: AEs were not collected for this trial
Arm/Group | Deep Inspiration Breath-hold (DIBH) Respiratory Motion
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-19): https://cdn.clinicaltrials.gov/large-docs/00/NCT04686500/Prot_SAP_000.pdf